CLINICAL TRIAL: NCT00275145
Title: Peripheral Effects of Exercise on Cardiovascular Health (STRRIDE II)
Brief Title: Effects of Resistance and Aerobic Exercise on Cardiovascular Health
Acronym: STRRIDE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00014514; R01HL057354 (NIH); 0438 (Other: Duke legacy IRB number)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2011-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Hyperlipidemia; Insulin Resistance; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Hyperlipidemias; Insulin Resistance; Metabolic Syndrome | interventions — Resistance Training; Exercise; carboxymethylmonobenzocyclooctyne

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Resistance Training (Experimental): 8 months of Resistance Exercise Training
  Interventions: Behavioral: Resistance Training
- Aerobic Exercise (Experimental): 8 months of Aerobic Exercise Training
  Interventions: Behavioral: Aerobic Exercise
- Combination RT & AT (Experimental): 8 months of Combined Aerobic and Resistance Exercise Training
  Interventions: Behavioral: Combo
- Control (Experimental): Control/sedentary intervention
  Interventions: Behavioral: Continued Sedentary lifestyle

INTERVENTIONS:
Behavioral: Resistance Training — Lifting weights 3 times per week; 8 different exercise each time; for each exercise, do three sets = lifting an appropriate weight between 8-12 for each set; rest 45 seconds (at least) between sets
  Arms: Resistance Training
Behavioral: Aerobic Exercise — Exercise at 75% of maximal capacity for approximately 2 hours per week
  Arms: Aerobic Exercise
Behavioral: Combo — Lift weights (as described in RT group) and do aerobic exercise (as described in Aerobic group
  Arms: Combination RT & AT
Behavioral: Continued Sedentary lifestyle — No changes
  Arms: Control

SUMMARY:
This study will investigate the separate and combined effects of aerobic and resistance training on cardiovascular risk factors in overweight men and women with mild to moderate dyslipidemia.

DETAILED DESCRIPTION:
BACKGROUND:

Substantial evidence supports a favorable relationship between cardiovascular fitness, physical activity, and cardiovascular health. In particular, it is well established that increased levels of physical activity result in favorable improvements in lipid and carbohydrate metabolism. There is also evidence that increased physical activity and cardiovascular fitness have beneficial effects on cardiovascular health, independent of the effects on specific cardiovascular risk factors. One hypothesis proposes that the beneficial effects of regular exercise in humans is mediated through peripheral mechanisms, in particular through the chronic adaptations in skeletal muscle to habitual exercise. The exercise exposure required to achieve health benefits is poorly defined and the mechanisms through which these beneficial adaptations occur are poorly understood. This study will investigate the peripheral biological mechanisms through which chronic physical activity alters carbohydrate metabolism and lipid metabolism, resulting in improvements in these parameters of cardiovascular health and fitness.

DESIGN NARRATIVE:

In Studies of a Targeted Risk Reduction Intervention through Defined Exercise II (STRRIDE II), participants will be randomly assigned to one of four exercise training regimens after a 4-month sedentary control period. After an initial ramp period of up to 2 months, participants will be asked to train for 6 months in a given exercise program. The programs differ either in the dose of aerobic exercise or in the mode (e.g., aerobic exercise, resistance exercise, or a combination). Parameters reflecting changes in carbohydrate and lipid metabolism will be studied at an integrative physiologic level and with measurable biological endpoints in peripheral skeletal muscle (capillary surface area). It is proposed that the elucidation of the peripheral mechanisms mediating the favorable responses in carbohydrate and lipid metabolism to chronic physical activity will lead to better understanding of the health benefits conferred by physical activity and cardiovascular fitness. This may also point the way toward better exercise recommendations for clients with significant cardiovascular risk factors. The purpose of this study is to investigate the peripheral biological mechanisms through which chronic physical activity will alter carbohydrate metabolism and lipid metabolism that results in improvement in parameters of cardiovascular health and fitness. The driving hypothesis is that the health benefits derived from habitual exercise are primarily mediated through adaptations occurring in skeletal muscle. The mechanism of change in skeletal muscle differs by the mode of exercise training. It is hypothesized that the health benefits of aerobic exercise are mediated primarily by qualitative changes in skeletal muscles (alterations in exposed capillary surface area in skeletal muscle induced by exercise training) and that the health benefits of resistance exercise are mediated primarily by quantitative changes in skeletal muscles (alterations in fiber area in skeletal muscle induced by exercise training). The investigators will use combination exercise regimens in moderately obese patients with mild to moderate lipid metabolic abnormalities in order to investigate whether induced alterations in skeletal muscle fiber area, metabolic capacity, and capillary surface area account for favorable alterations in insulin sensitivity, glucose metabolism, lipoprotein levels, and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (exercises fewer than two times per week)
* Overweight or mildly obese (body mass index [BMI] of 25 to 35 kg/m2) with mild to moderate lipid abnormalities (either LDL cholesterol 130 to 190 mg/dl or HDL cholesterol less than 40 mg/dl for men or 5 less than 45 mg/dl for women)

Exclusion Criteria:

* Diabetes
* Hypertension
* Other metabolic or musculoskeletal diseases
* Current use of or intent to diet
* Use of confounding medication
* Overt presence of coronary heart disease
* Unwilling to be randomized to any group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Major Cardiometabolic Risk Factors: lipoproteins; Ectopic Fat (Visceral Fat, Liver fat); body composition (fat mass, lean body mass; and Insulin Sensitivity | Month 0, Month 4, Year 1, and Year 1 plus 2 weeks

SECONDARY OUTCOMES:
Metabolic Syndrome (ATP III defined); Maximal Oxygen consumption; muscle biopsy measures (oxidative enzymes, capillary density, myofiber diameter) | 0 mths, 4 mths, 1 year and 1 year and 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William E. Kraus, Study Chair — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Jiang R, Collins KA, Huffman KM, Hauser ER, Hubal MJ, Johnson JL, Williams RB, Siegler IC, Kraus WE. Genome-Wide Genetic Analysis of Dropout in a Controlled Exercise Intervention in Sedentary Adults With Overweight or Obesity and Cardiometabolic Disease. Ann Behav Med. 2024 Apr 11;58(5):363-374. doi: 10.1093/abm/kaae011. PMID 38489667
- [Derived] Collins KA, Fos LB, Ross LM, Slentz CA, Davis PG, Willis LH, Piner LW, Bateman LA, Houmard JA, Kraus WE. Aerobic, Resistance, and Combination Training on Health-Related Quality of Life: The STRRIDE-AT/RT Randomized Trial. Front Sports Act Living. 2021 Feb 11;2:620300. doi: 10.3389/fspor.2020.620300. eCollection 2020. PMID 33644749
- [Derived] AbouAssi H, Slentz CA, Mikus CR, Tanner CJ, Bateman LA, Willis LH, Shields AT, Piner LW, Penry LE, Kraus EA, Huffman KM, Bales CW, Houmard JA, Kraus WE. The effects of aerobic, resistance, and combination training on insulin sensitivity and secretion in overweight adults from STRRIDE AT/RT: a randomized trial. J Appl Physiol (1985). 2015 Jun 15;118(12):1474-82. doi: 10.1152/japplphysiol.00509.2014. PMID 25882384
- [Derived] Moker EA, Bateman LA, Kraus WE, Pescatello LS. The relationship between the blood pressure responses to exercise following training and detraining periods. PLoS One. 2014 Sep 10;9(9):e105755. doi: 10.1371/journal.pone.0105755. eCollection 2014. PMID 25208075
- [Derived] Huffman KM, Koves TR, Hubal MJ, Abouassi H, Beri N, Bateman LA, Stevens RD, Ilkayeva OR, Hoffman EP, Muoio DM, Kraus WE. Metabolite signatures of exercise training in human skeletal muscle relate to mitochondrial remodelling and cardiometabolic fitness. Diabetologia. 2014 Nov;57(11):2282-95. doi: 10.1007/s00125-014-3343-4. Epub 2014 Aug 5. PMID 25091629
- [Derived] Willis LH, Slentz CA, Bateman LA, Shields AT, Piner LW, Bales CW, Houmard JA, Kraus WE. Effects of aerobic and/or resistance training on body mass and fat mass in overweight or obese adults. J Appl Physiol (1985). 2012 Dec 15;113(12):1831-7. doi: 10.1152/japplphysiol.01370.2011. Epub 2012 Sep 27. PMID 23019316
- [Derived] Slentz CA, Bateman LA, Willis LH, Shields AT, Tanner CJ, Piner LW, Hawk VH, Muehlbauer MJ, Samsa GP, Nelson RC, Huffman KM, Bales CW, Houmard JA, Kraus WE. Effects of aerobic vs. resistance training on visceral and liver fat stores, liver enzymes, and insulin resistance by HOMA in overweight adults from STRRIDE AT/RT. Am J Physiol Endocrinol Metab. 2011 Nov;301(5):E1033-9. doi: 10.1152/ajpendo.00291.2011. Epub 2011 Aug 16. PMID 21846904
- [Derived] Bateman LA, Slentz CA, Willis LH, Shields AT, Piner LW, Bales CW, Houmard JA, Kraus WE. Comparison of aerobic versus resistance exercise training effects on metabolic syndrome (from the Studies of a Targeted Risk Reduction Intervention Through Defined Exercise - STRRIDE-AT/RT). Am J Cardiol. 2011 Sep 15;108(6):838-44. doi: 10.1016/j.amjcard.2011.04.037. Epub 2011 Jul 7. PMID 21741606